CLINICAL TRIAL: NCT01793246
Title: Registry Trial to Determine pCLE Image Interpretation Criteria and Preliminary Accuracy: Discrete Pulmonary Lesions and Acute Rejection in Transplanted Lungs
Brief Title: Registry Trial to Determine pCLE Image Interpretation Criteria and Preliminary Accuracy in the Lung
Acronym: BREATH
Status: Completed | Type: Observational
Sponsor: Mauna Kea Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: MKT_2012_lung_01
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Lung Neoplasms; Disorder Related to Lung Transplantation
Keywords: lung cancer; lung neoplasms; lung transplant
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pCLE for Discrete lung lesions: Patients undergoing bronchoscopy for the diagnosis of a lesion with probe based laser endomicroscopy (pCLE) imaging before biopsy
  Interventions: Device: probe based laser endomicroscopy (pCLE)
- pCLE for acute lung transplant rejection: Patients undergoing bronchoscopy for the detection of acute rejection of lung transplant with probe based laser endomicroscopy (pCLE) imaging before biopsy
  Interventions: Device: probe based laser endomicroscopy (pCLE)

INTERVENTIONS:
Device: probe based laser endomicroscopy (pCLE) — pCLE will be added to standard bronchoscopy for the purpose of characterizing lung cancer or for characterizing of acute rejection in transplanted lungs.
  Other Names: Cellvizio; pCLE; probe based confocal laser endomicroscopy; optical biopsy; optical endomicroscopy

SUMMARY:
Patients will be enrolled that are undergoing bronchoscopy for diagnosis of discrete lung lesions or for detection of acute rejection following lung transplants. The hypothesis is that bronchoscopy together with probe-based endomicroscopy (pCLE)results in improved and/or incremental diagnostic yield (definitive diagnosis) over conventional bronchoscopy.

DETAILED DESCRIPTION:
The primary aim of this study is to develop the criteria to differentiate healthy versus diseased tissue in patient with discrete lung lesions or to characterize acute lung rejection in patients with transplanted lungs. Once these criteria have been defined, the diagnostic parameters and the reproducibility of pCLE will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years of age
* Willing and able to comply with study procedures and provide written informed consent to participate in the study
* Indeterminate discrete nodule(s) suspicious for cancer scheduled for diagnostic bronchoscopy
* Newly discovered &/or prior discovered non classified nodules, hard to define based on CT scan
* Purpose of bronchoscopy is for diagnosis of lesion(s) - can be solitary pulmonary nodule or multiple lesions
* All lesion locations are acceptable
* Any patient undergoing clinically indicated bronchoscopies after lung transplantation
* Patients post transplant showing clinical signs of acute rejection >3 weeks; < 1 year
* Patient with single or double lung transplant

Exclusion Criteria:

* Contraindication to short-acting anesthetic agents;
* Contraindications to transbronchial biopsy
* Bleeding diathesis;
* A pacemaker/defibrillator;
* A diagnosis by other means (sputum cytology, microbiology).
* Unwilling To Consent
* Unable To Safely Tolerate A Bronchoscopic Procedure
* Unwilling To Comply With Surveillance Bronchoscopy Follow Up
* Chronic Rejection
* Fungal Disease
* Ax Histological Assessment Or Incomplete Biopsy Procedure Should Be Considered As A Screen Failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are 18 years of age or older with a clinical indication for a Bronchoscopic procedure for:
  * Discrete Lung Lesions
  * Surveillance or Symptoms of Acute Rejection in Lung Transplants
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2013-02; Primary Completion 2016-12-24 (Actual); Study Completion 2016-12-24 (Actual)

PRIMARY OUTCOMES:
Development of criteria for the characterization of discrete lung lesions and for characterization of acute lung rejection in lung transplant. | Up to 12 months
  For Group 1 - Discrete lung lesions
Diagnostic performance of the pCLE image interpretation criteria for discrete lung lesions and for acute lung rejection in lung transplant. | Up to 12 months.
  For Group 2 - Transplant rejection

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Keller, MD, Principal Investigator — Mayo Clinic; Kyle Hogarth, MD, Principal Investigator — University of Chicago; Doug Arenberg, MD, Principal Investigator — University of Michigan; Adam Wellikoff, MD, Principal Investigator — Louisiana State University Health Sciences Center Shreveport
Locations (9):
- United States (9):
  - St. Joseph's Medical Center, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - Columbus Regional Hospital, Columbus, Indiana
  - University of Louisiana Shreveport, Shreveport, Louisiana
  - Walter Reed Military Medical Center, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Rochester, Rochester, New York
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Background] Meining A, Chen YK, Pleskow D, Stevens P, Shah RJ, Chuttani R, Michalek J, Slivka A. Direct visualization of indeterminate pancreaticobiliary strictures with probe-based confocal laser endomicroscopy: a multicenter experience. Gastrointest Endosc. 2011 Nov;74(5):961-8. doi: 10.1016/j.gie.2011.05.009. Epub 2011 Jul 29. PMID 21802675
- [Background] Sharma P, Meining AR, Coron E, Lightdale CJ, Wolfsen HC, Bansal A, Bajbouj M, Galmiche JP, Abrams JA, Rastogi A, Gupta N, Michalek JE, Lauwers GY, Wallace MB. Real-time increased detection of neoplastic tissue in Barrett's esophagus with probe-based confocal laser endomicroscopy: final results of an international multicenter, prospective, randomized, controlled trial. Gastrointest Endosc. 2011 Sep;74(3):465-72. doi: 10.1016/j.gie.2011.04.004. Epub 2011 Jul 13. PMID 21741642
- [Background] Pohl H, Rosch T, Vieth M, Koch M, Becker V, Anders M, Khalifa AC, Meining A. Miniprobe confocal laser microscopy for the detection of invisible neoplasia in patients with Barrett's oesophagus. Gut. 2008 Dec;57(12):1648-53. doi: 10.1136/gut.2008.157461. Epub 2008 Aug 28. PMID 18755886
- [Background] Newton RC, Kemp SV, Yang GZ, Elson DS, Darzi A, Shah PL. Imaging parenchymal lung diseases with confocal endomicroscopy. Respir Med. 2012 Jan;106(1):127-37. doi: 10.1016/j.rmed.2011.09.009. Epub 2011 Oct 14. PMID 22000588
- [Background] Yick CY, von der Thusen JH, Bel EH, Sterk PJ, Kunst PW. In vivo imaging of the airway wall in asthma: fibered confocal fluorescence microscopy in relation to histology and lung function. Respir Res. 2011 Jun 23;12(1):85. doi: 10.1186/1465-9921-12-85. PMID 21699692
- [Background] Thiberville L, Salaun M, Lachkar S, Dominique S, Moreno-Swirc S, Vever-Bizet C, Bourg-Heckly G. Human in vivo fluorescence microimaging of the alveolar ducts and sacs during bronchoscopy. Eur Respir J. 2009 May;33(5):974-85. doi: 10.1183/09031936.00083708. Epub 2009 Feb 12. PMID 19213792
- [Background] Henschke CI, Naidich DP, Yankelevitz DF, McGuinness G, McCauley DI, Smith JP, Libby D, Pasmantier M, Vazquez M, Koizumi J, Flieder D, Altorki N, Miettinen OS. Early lung cancer action project: initial findings on repeat screenings. Cancer. 2001 Jul 1;92(1):153-9. doi: 10.1002/1097-0142(20010701)92:13.0.co;2-s. PMID 11443621
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Ikeda N, Hayashi A, Iwasaki K, Honda H, Tsuboi M, Usuda J, Kato H. Comprehensive diagnostic bronchoscopy of central type early stage lung cancer. Lung Cancer. 2007 Jun;56(3):295-302. doi: 10.1016/j.lungcan.2007.01.009. Epub 2007 Feb 8. PMID 17291623
- [Background] Wang Memoli JS, Nietert PJ, Silvestri GA. Meta-analysis of guided bronchoscopy for the evaluation of the pulmonary nodule. Chest. 2012 Aug;142(2):385-393. doi: 10.1378/chest.11-1764. PMID 21980059
- [Background] Gildea TR, Mazzone PJ, Karnak D, Meziane M, Mehta AC. Electromagnetic navigation diagnostic bronchoscopy: a prospective study. Am J Respir Crit Care Med. 2006 Nov 1;174(9):982-9. doi: 10.1164/rccm.200603-344OC. Epub 2006 Jul 27. PMID 16873767
- [Background] Wilson DS, Bartlett RJ. Improved Diagnostic Yield of Bronchoscopy in a Community Practice: Combination of Electromagnetic Navigation System and Rapid On-site Evaluation. Journal of Bronchology & Interventional Pulmonology 2007;14:227-232 10.1097/LBR.0b013e31815a7b00.
- [Background] Ohtani K, Lee AM, Lam S. Frontiers in bronchoscopic imaging. Respirology. 2012 Feb;17(2):261-9. doi: 10.1111/j.1440-1843.2011.02108.x. PMID 22126413
- [Background] Salaun M, Bourg-Heckly G, Thiberville L. [Confocal endomicroscopy of the lung: from the bronchus to the alveolus]. Rev Mal Respir. 2010 Jun;27(6):579-88. doi: 10.1016/j.rmr.2009.12.009. Epub 2010 Jun 2. French. PMID 20610073
- [Background] Thiberville L, Salaun M. Bronchoscopic advances: on the way to the cells. Respiration. 2010;79(6):441-9. doi: 10.1159/000313495. Epub 2010 May 12. PMID 20431326
- [Background] Filner JJ, Bonura EJ, Lau ST, Abounasr KK, Naidich D, Morice RC, Eapen GA, Jimenez CA, Casal RF, Ost D. Bronchoscopic fibered confocal fluorescence microscopy image characteristics and pathologic correlations. J Bronchology Interv Pulmonol. 2011 Jan;18(1):23-30. doi: 10.1097/LBR.0b013e318203da1c. PMID 23169014
- [Background] DeVito Dabbs A, Hoffman LA, Iacono AT, Wells CL, Grgurich W, Zullo TG, McCurry KR, Dauber JH. Pattern and predictors of early rejection after lung transplantation. Am J Crit Care. 2003 Nov;12(6):497-507. PMID 14619355
- [Background] Gotway MB, Dawn SK, Sellami D, Golden JA, Reddy GP, Keith FM, Webb WR. Acute rejection following lung transplantation: limitations in accuracy of thin-section CT for diagnosis. Radiology. 2001 Oct;221(1):207-12. doi: 10.1148/radiol.2211010380. PMID 11568342
- [Background] MacMahon H, Austin JH, Gamsu G, Herold CJ, Jett JR, Naidich DP, Patz EF Jr, Swensen SJ; Fleischner Society. Guidelines for management of small pulmonary nodules detected on CT scans: a statement from the Fleischner Society. Radiology. 2005 Nov;237(2):395-400. doi: 10.1148/radiol.2372041887. PMID 16244247